CLINICAL TRIAL: NCT03658005
Title: Population-Based Pharmacokinetic / Pharmacodynamic Modeling of the Effect of Free Ticagrelor Fraction on the Platelet Membrane in Post Myocardial Infarction Patients
Brief Title: Effect of Free Ticagrelor Fraction on Platelet Membrane Post MI
Acronym: PLATIME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/371
Record Dates: First submitted 2018-07-12; First posted 2018-09-05 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Ticagrelor; acute coronary syndrome; anti-platelet drug
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Adult (>18 years, <90 years) patients admitted and treated for acute myocardial infarction, and whose treatment includes ticagrelor in association with aspirin.
  Blood samples will be taken at 3 timepoints between two doses of ticagrelor (taken at 12 hours interval).
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — 3 blood samples, for a maximum of 60mL, will be taken at 0-3h, 3-6h and >6h, between two doses of ticagrelor (taken at 0 and 12 hours).

SUMMARY:
The purpose of this study is to assess:

* the population pharmacokinetics of unbound ticagrelor and its metabolite in acute coronary syndrome patients treated by ticagrelor
* ticagrelor and its metabolite levels by LC-MS/MS

DETAILED DESCRIPTION:
Ticagrelor is an anti-platelet agent of the cyclopentyltriazolopyrimidine class. It is administered by the oral route, rapidly absorbed (2-3 hours), and has a bio-availability estimated at around 36%. Contrary to other P2Y12 inhibitors, ticagrelor is not a pro-drug and does not need to be metabolized to exert is pharmacodynamic effect. It had been previously showed that stimulation of platelets by ADP or inhibitors of platelets by ticagrelor modified the organisation of the platelet membrane, with a re-distribution of cholesterol and P2Y12 receptors towards the lipid rafts. This suggests that lipid membranes and cholesterol may play an important role in the anti-platelet activity of ticagrelor.

In this context, the aim of the study is to assess:

* the population pharmacokinetics of unbound ticagrelor and its metabolite in acute coronary syndrome patients treated by ticagrelor
* ticagrelor and its metabolite levels by LC-MS/MS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years and less than 90 years,
* Patients admitted for myocardial infarction treated with ticagrelor in association with aspirin.
* Patients affiliated to a social security system (or be a beneficiary thereof);
* Sign written informed consent indicating that they have understood the study procedures and objectives, and that they accept to participate and adhere to the study requirements.

Exclusion Criteria:

* Patients with limited legal capacity or patients under legal guardianship
* Patients under judicial protection
* Patients not affiliated to any social security system
* Patients taking any antiplatelet agent other than ticagrelor Patients taking ticagrelor for <48 hours (treatment not stabilised) Patients with hemoglobin concentration <10 g/dL on the most recent blood test

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Cardiology department with a main diagnosis of acute coronary syndrome and treated with a treatment combination including ticagrelor and aspirin.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-04-09 (Estimated); Study Completion 2022-04-09 (Estimated)

PRIMARY OUTCOMES:
concentration of unbound ticagrelor and its metabolite | at 3 hours after administration of the first dose of ticagrelor
  Concentration of unbound ticagrelor and its active metabolite in acute coronary syndrome patients treated by ticagrelor and aspirin
concentration of unbound ticagrelor and its metabolite | at 6 hours after administration of the first dose of ticagrelor
  Concentration of unbound ticagrelor and its active metabolite in acute coronary syndrome patients treated by ticagrelor and aspirin
concentration of unbound ticagrelor and its metabolite | at 12 hours after administration of the first dose of ticagrelor
  Concentration of unbound ticagrelor and its active metabolite in acute coronary syndrome patients treated by ticagrelor and aspirin

SECONDARY OUTCOMES:
Assess the method of determination of ticagrelor concentration | at 3 hours after administration of the first dose of ticagrelor
  Identify the optimum settings for the measurement of the concentration of ticagrelor (total and free fraction) and its active metabolite in the plasma by LC-MS/MS
Assess the method of determination of ticagrelor concentration | at 6 hours after administration of the first dose of ticagrelor
  Identify the optimum settings for the measurement of the concentration of ticagrelor (total and free fraction) and its active metabolite in the plasma by LC-MS/MS
Assess the method of determination of ticagrelor concentration | at 12 hours after administration of the first dose of ticagrelor
  Identify the optimum settings for the measurement of the concentration of ticagrelor (total and free fraction) and its active metabolite in the plasma by LC-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Meneveau, MD, PhD, Principal Investigator — Dept of Cardiology, CHU Besancon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No